CLINICAL TRIAL: NCT05693116
Title: Survival and Prognostic Factors of Squamous Cell Carcinoma of the Nasal Vestibule: a Multi-centre Study
Brief Title: Survival and Prognostic Factors of Squamous Cell Carcinoma of the Nasal Vestibule
Acronym: NV-SCC
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 3273
Record Dates: First submitted 2022-12-08; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Nasal Vestibule Carcinoma; Rhinectomy; Nasal Vestibule; Squamous Cell Carcinoma
Keywords: nasal vestibule; squamous cell carcinoma; rhinectomy
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nasal Vestibule Squamous Cell Carcinoma: Patients affected by primary squamous cell carcinoma of the nasal vestibule. Patients will be treated with upfront surgery according to the current practice and followed to identify any possible factor affecting prognosis.
  Interventions: Procedure: Rhinectomy

INTERVENTIONS:
Procedure: Rhinectomy — Surgery will be performed according to extension of the tumour, i.e. local resection limited to the vestibule, partial rhinectomy, total rhinectomy, extended total rhinectomy

SUMMARY:
The goal of this observational study is to learn about survival and prognostic factors in patients who underwent surgical treatment for primary squamous cell carcinoma of the nasal vestibule. The main questions it aims to answer are:

* what is the prognosis of patients affected by squamous cell carcinoma of the nasal vestibule?
* are there any specific factors that could influence prognosis?
* is it possible to elaborate a new staging system, able to overcome the limitations of the currently used ones? Data about patients, tumour and type of surgery performed will be collected. Participants will be followed-up for a minimum 6 months period after surgery.

DETAILED DESCRIPTION:
This study will address the survival of patients with squamous cell carcinoma of the nasal vestibule (NV-SCC), and it will analyze factors influencing it.

In particular, apart from demographic features of the patient, data regarding the origin of the tumour and its extension will be collected and the lesion will be restaged according the the three classification systems used at present (Wang's classification, AJCC for nasal cavity cancers, AJCC for non-melanomatous skin cancer of head and neck region), given the current controversy regarding the best staging system. Furthermore data related to the surgery and the final histology will be collected.

All collected data will be analyzed in order to investigate any possible factor related to overall survival, disease specific survival and disease free survival.

Patients will be followed for a minimum of 6 months up to 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of squamous cell carcinoma of the nasal vestibule
* underwent upfront surgical treatment with curative intent
* availability of clinical and radiological data for cT reassessment
* availability of histological samples for pT reassessment
* follow-up of at least 6 months after surgery.

Exclusion Criteria:

* patients initially referred for disease persistence or recurrence
* patients affected by tumour involving the nasal vestibule but originating from other sites (eg. nasal cavities, skin of the nasal pyramid or upper lip)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by primary squamous cell carcinoma of the nasal vestibule.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Survival | From time of enrollment to event (death, recurrence) up to 60 months.
  Overall Survival
Survival | From time of enrollment to event (death, recurrence) up to 60 months.
  Disease Free Survival
Survival | From time of enrollment to event (death, recurrence) up to 60 months.
  Disease Specific Survival

SECONDARY OUTCOMES:
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Gender
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Age
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Site of origin of the tumour
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Subsites involved by the tumour
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  cT stage (according to TNM nasal cavities, Wang classification, TNM skin)
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  cN stage
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  pT stage (according to TNM nasal cavities, Wang classification, TNM skin)
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  pN stage (according to TNM nasal cavities, Wang classification, TNM skin)
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Grade
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Dimensions
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Depth of infiltration
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Perineural invasion
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Perivascular invasion
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Surgical margin status
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Surgical procedure
Factors influencing survival (demographics, tumour-related, surgery-related) | From time of enrollment to event (death, recurrence) up to 60 months.
  Adjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ferreli, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (6):
- Centre Hospitalier Universitaire de Toulouse, Toulouse, Touluse, France
- Italy (4):
  - Humanitas Research Hospital, Rozzano, Milan
  - Cagliari University Hospital, Cagliari
  - IRCCS San Raffaele Hospital, Milan
  - Varese University Hospital, Varese
- Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreli F, Pirola F, Di Santo D, De Virgilio A, Spriano G, Mercante G. A critical analysis of the classifications of squamous cell carcinoma of the nasal vestibule. Oral Oncol. 2022 Jun;129:105880. doi: 10.1016/j.oraloncology.2022.105880. Epub 2022 Apr 28. No abstract available. PMID 35490569
- [Background] Lambertoni A, Cherubino M, Battaglia P, De Col A, Giovannardi M, Antognoni P, Valdatta L, Karligkiotis A, Bignami M, Castelnuovo P, Turri-Zanoni M. Squamous Cell Carcinoma of Nasal Vestibule and Pyramid: Outcomes and Reconstructive Strategies. Laryngoscope. 2021 Apr;131(4):E1198-E1208. doi: 10.1002/lary.29107. Epub 2020 Oct 2. PMID 33006408
- [Background] Chabrillac E, Talawdekar A, Garikipati S, Varley I, Sionis S, Beasley N, Jackson R. A single centre's experience of 23 cases of total rhinectomy for the treatment of squamous cell carcinoma involving the nasal vestibule. Eur Arch Otorhinolaryngol. 2022 Apr;279(4):2069-2075. doi: 10.1007/s00405-021-06972-6. Epub 2021 Jul 5. PMID 34223976